CLINICAL TRIAL: NCT04476303
Title: A Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Phase I Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetics of BEY2153 After Oral Administration in Healthy Young and Elderly Male Volunteers.
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of BEY2153 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeyondBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BEY-2019-01
Record Dates: First submitted 2020-07-13; First posted 2020-07-20 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SAD (#6 Cohort) (Experimental): Drug: BEY2153 or placebo subjects will receive single ascending dose of BEY2153 or placebo once.
  Interventions: Drug: BEY2153
- SAD (#1 Cohort) - Food effect evaluation (Experimental): Drug: BEY2153 or placebo subjects will receive single ascending dose of BEY2153 or placebo for two periods at 7 days interval, with both fasting and after high fat meal.
  Interventions: Drug: BEY2153
- MAD (#4 Cohort) (Experimental): Drug: BEY2153 or placebo subjects will receive multiple ascending dose of BEY2153 or placebo for 7 days.
  Interventions: Drug: BEY2153

INTERVENTIONS:
Drug: BEY2153 — Capsule

SUMMARY:
This is a first in human Phase 1 study to evaluate the safety, tolerability and pharmacokinetics with healthy young and elderly adult male volunteers after receiving single and multiple ascending dose of BEY2153.

DETAILED DESCRIPTION:
Healthy young and elderly adult volunteers who meet the criteria, will be treated single and multiple ascending dose of BEY2153 or placebo orally. Food effect evaluation study will be conducted with single ascending dose. After the single ascending dose study, independent external experts will review blinded data and multiple ascending dose study will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Young adult: A healthy Korean male aged 19 to 45 (inclusive) years at the time of screening Elderly adult: A healthy Korean male aged over 65 (inclusive) years at the time of screening"
2. Subjects weighing between 55 kg and 90 kg with BMI between 18.0 and 27.0 kg/m2 (inclusive) at screening.
3. Subjects who have listened to the detailed description of this clinical trial and have fully understood, and who have agreed in writing to voluntarily participate and observe the precautions prior to receiving any of the screening procedures
4. Subjects who is eligible for this clinical trial by the investigator's judgement with laboratory test results and physical-examination findings and etc.

Exclusion Criteria:

1. Young adult / Elderly adult: Subjects with evidence or a history of clinically significant hepatic, renal, neurologic, immunologic, pulmonary, endocrine or hematological, neoplastic, cardiovascular, psychiatric diseases (mood disorder, obsessive-compulsive disorder etc.).
2. Subjects with evidence or a history of gastrointestinal disease or with history of gastrointestinal surgery that may affect assessment of safety, PK characteristics of study drug.
3. Subjects who showed significant abnormalities at neurologic examination at screening visit.
4. Subjects who showed any abnormalities at vital signs
5. Subjects who showed any abnormalities at blood test
6. Subjects with serum AST (SGOT) or ALT (SGPT) level or total bilirubin exceed 1.5 times the upper limit of the normal range at screening
7. Subjects who showed any abnormalities at ECG subsection
8. Subjects who are hypersensitive to drugs, or who have clinically significant hypersensitivity reactions history.
9. Subjects with a history of alcohol or drug abuse or subjects who showed positive results for abuse drug at urine drug screening test.
10. Subjects who consume alcohol continuously or who are unable to abstain from drinking from the time of consent until the end of the clinical trial.
11. Smokers
12. Subjects who had recessive disease, symptomatic infection, virus, bacteria or fungus infection 1 week before the first study drug administration.
13. Subjects who have taken any prescribed drug or herbal medicine within two weeks prior to the first study drug administration. Non-prescribed medicine (OTC) or vitamin supplement prohibit within one week prior to the first study drug administration or subjects whose administrations are predicted.
14. Subjects who have participated and taken investigational drug in any other clinical trial within six months prior to study drug administration
15. Subjects who showed positive result for HBs antigen, HCV antibody, HIV antigen-antibody test at screening
16. Subjects who had whole blood donation, apheresis or blood transfusion within 3 months before the first study drug administration.
17. Subjects who had grapefruit containing food from 3 days before the scheduled date of the first study drug administration to discharge and those who cannot be prevented from taking it during the study period.
18. Subjects who consume or are unable to abstain from products containing caffeine from 3 days before the scheduled date of the first study drug administration to discharge, and those who cannot be prevented from taking it during the study period.
19. Subjects who do not agree to use following medically appropriate method of contraception and not to donate sperm starting from subject enrollment to 90 days after last administration of investigational product.
20. Subjects judged ineligible for the study after a review of the clinical laboratory results by the investigator or for other reasons.

Ages: 19 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Day 1 to Day 9
Area Under the Curve (AUC) | Day 1 to Day 9
Apparent terminal elimination half-life (t1/2) | Day 1 to Day 9
Apparent clearance (CL/F) | Day 1 to Day 9
Apparent volume of distribution (Vz/F) | Day 1 to Day 9

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 48 days
Incidence of Serious Adverse Events (SAEs) | Up to 48 days
Incidence of clinically significant changes in vital signs | Up to 18 days
Incidence of clinically significant changes in 12-Lead electrocardiogram (ECG) parameters | Up to 18 days
Incidence of clinically significant changes in clinical laboratory results | Up to 18 days
Incidence of clinically significant changes in physical examination | Up to 18 days

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No